CLINICAL TRIAL: NCT02793479
Title: National Registry for Radiofrequency Ablation in Patients With Barrett's Esophagus
Brief Title: Radiofrequency Ablation in Patients With Barrett's Esophagus
Acronym: RABE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Matthias Paireder (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor-Investigator, Matthias Paireder, Medical Doctor, Austrian Society Of Surgical Oncology
Organization: Austrian Society Of Surgical Oncology (Other)
Other Study IDs: AUT-RFA-Registry-01
Record Dates: First submitted 2016-06-01; First posted 2016-06-08 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Barrett's Esophagus; Radiofrequency Ablation; Gastroesophageal Reflux Disease
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years

GROUPS / COHORTS (1):
- BE: Patients presenting Barrett's Esophagus as a complication of a gastroesophageal reflux disease.

SUMMARY:
The aim of this study is to establish a nationwide registry to collect data regarding the treatment of Barrett's Esophagus (BE) with radiofrequency ablation. The objective of this registry is to increase the number of data and therefore obtain a raise of quality assurance and improve outcome and patient security. Furthermore to provide participating physicians information and experience for treatment details in the therapy of BE.

DETAILED DESCRIPTION:
For treatment of Barrett's Esophagus (BE), a condition considered as a complication of the gastroesophageal reflux disease (GERD), radiofrequency ablation (RFA) was introduced as a new method over 10 years ago. This method is already established in treating low- and high-grade dysplastic BE, but there is also a recommendation in therapy of non-dysplastic Barrett's esophagus (NDBE), if patients provide a increased cancer risk profile, such as long history of GERD (over 10 years), large hiatal hernia (over 3cm), esophagitis, history of BE with dysplasia or positive family history for gastrointestinal cancer.

In Austria 1 - 3% of the population is estimated to develop BE. The treatment numbers in each specialized centers therefore is low. To guarantee a better and more potent data analysis, the establishment of a nationwide registry is crucial. Furthermore this is essential to raise quality assurance and improve outcome and patients will benefit eventually.

The aim is the participation of about 10 departments, which are all qualified centers and experts, who offer RFA as a treatment for BE. Thus data can be collected and interpreted more exact due to the increased number of treated patients. For the purpose of data collection a structured electronic form will be used. This will further improve treatment documentation and quality.

Documentation will be performed in participating local centers. High priority is patient safety and data de-personalization. Data administration and data input should be performed through qualified medical personal via an online documentation platform. Original patients charts are archived at each center and data de-personalization is guaranteed via consecutive numbering when submitted to the study center.

Therefore protection of privacy of participating patients can be assured.

The registry should contain basis data of the patient as well as specific treatment data.

1. Patient data Personal identification number (PIN) Sex Age Place of residence - county
2. GERD history Typical, atypical symptoms Leading symptom Since when symptomatically Since when proton-pump inhibitor (PPI) treatment, dose Fundoplication y/n, Type, Date
3. Endoscopy Date of diagnosis - Date of endoscopy Endoscopic Classification (Prague) Histological Classification
4. Treatment Data Catheter type: 360°, 90° Energy: 10/12 J/cm2 Ablation catheter 18, 22, 25, 28, 31mm Ablation from … to … ab ore, length Complications
5. Follow Up Date Endoscopic Classification (Prague) Histological Classification Complete remission of intestinal metaplasia (CR-IM) Proton-pump inhibitor (PPI), Dose

Inclusion of 500 patients a study period of two years is planned. There will be a possible extension of the study period, if the registry is successful.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histological confirmed BE, who give their informed consent for participation in an anonymized registry.

Exclusion Criteria:

* Patients, who do not give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each center should define a system for identification and eligibility screening of patients.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients treated with Radiofrequency Ablation for Barrett's Esophagus in Austria | 5 years
Elimination Rate of Barrett's Esophagus in the study population | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian F Schoppmann, MD, Study Director — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Chandrasoma P, Makarewicz K, Wickramasinghe K, Ma Y, Demeester T. A proposal for a new validated histological definition of the gastroesophageal junction. Hum Pathol. 2006 Jan;37(1):40-7. doi: 10.1016/j.humpath.2005.09.019. Epub 2005 Nov 28. PMID 16360414
- [Background] Fleischer DE, Odze R, Overholt BF, Carroll J, Chang KJ, Das A, Goldblum J, Miller D, Lightdale CJ, Peters J, Rothstein R, Sharma VK, Smith D, Velanovich V, Wolfsen H, Triadafilopoulos G. The case for endoscopic treatment of non-dysplastic and low-grade dysplastic Barrett's esophagus. Dig Dis Sci. 2010 Jul;55(7):1918-31. doi: 10.1007/s10620-010-1218-1. Epub 2010 Apr 20. PMID 20405211
- [Background] Fleischer DE, Overholt BF, Sharma VK, Reymunde A, Kimmey MB, Chuttani R, Chang KJ, Muthasamy R, Lightdale CJ, Santiago N, Pleskow DK, Dean PJ, Wang KK. Endoscopic radiofrequency ablation for Barrett's esophagus: 5-year outcomes from a prospective multicenter trial. Endoscopy. 2010 Oct;42(10):781-9. doi: 10.1055/s-0030-1255779. Epub 2010 Sep 20. PMID 20857372